CLINICAL TRIAL: NCT02021864
Title: Effect of Treatment of Vitamin D Deficiency During Pregnancy on Hypocalcemia
Brief Title: Vitamin D Treatment and Hypocalcemic Pregnant Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Sima Hashemipour (Other)
Responsible Party: Sponsor-Investigator, Dr. Sima Hashemipour, assistant professor of endocrinology and metabolism, Sina Hospital, Iran
Organization: Sina Hospital, Iran (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: hypocalcemia of pregnancy
Record Dates: First submitted 2013-12-20; First posted 2013-12-27 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Pregnancy Complications
Keywords: hypocalcemia, pregnancy, vitamin D
MeSH Terms: conditions — Pregnancy Complications; Hypocalcemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vitamin D3, prenatal multivitamin (Experimental): vitamin D3 50,000 unit/week for 8 weeks, daily prenatal multivitamin containing elemental calcium 250 mg/day and vitamin D3 400 unit
  Interventions: Drug: vitamin D3 50,000 unit; Drug: prenatal multivitamin
- prenatal multivitamin (Active Comparator): daily prenatal multivitamin containing elemental calcium 250 mg/day and vitamin D3 400 unit
  Interventions: Drug: prenatal multivitamin

INTERVENTIONS:
Drug: vitamin D3 50,000 unit — vitamin D3 50,000 unit/week for 8 weeks
  Arms: vitamin D3, prenatal multivitamin
Drug: prenatal multivitamin — daily prenatal multivitamin containing elemental calcium 250 mg/day and vitamin D3 400 unit

SUMMARY:
* Pregnant women in 24-26 gestational week will be recruited.Serum calcium and 25(OH)D will be evaluated and women with mild hypocalcemia (serum calcium 8-8.6 mg/dl) and 25(OH)D less than 30ng/ml will be entered to study. .
* Excluding criteria are: gestational diabetes or diabetes before pregnancy, severe preeclampsia, chronic hypertension, fetal anomaly, oligohydramnios or polyhydramnios, parathyroid disorders, hepatic or renal diseases, malnutrition , use of anti- convulsive and immunosuppressive drugs.
* Participants will randomly assigned in to two groups of intervention and control groups .Randomization will be done by random number generator. Intervention group will receive weekly vitamin D3, 50,000 unit for 8 weeks plus daily prenatal multivitamin containing elemental calcium 250 mg/day and vitamin D3 400 unit , control group will receive daily prenatal multivitamin.
* At the time of delivery, serum calcium, 25(OH)D of mothers, maternal weight gain during study , Serum calcium and 25(OH)D of newborns and neonatal growth indices ( length, weight, head circumference ) will be compared between two groups.

ELIGIBILITY:
Inclusion Criteria:

gestational age of 24-26weeks,mild hypocalcemia (ca=8-8.6mg/dl),singleton pregnancy, body mass index (BMI) of 19-26 -

Exclusion Criteria:

moderate to sever hypocalcemia(ca<8mg/dl), gestational diabetes or diabetes before pregnancy, severe preeclampsia, chronic hypertension, fetal anomaly, oligohydramnios or polyhydramnios, parathyroid disorders, hepatic or renal diseases, malnutrition , use of anti- convulsive and immunosuppressive drugs

-

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
percentage of hypocalcemic subjects at the ens of study | 12-14 weeks
  women in 24-26 weeks of pregnancy will be enrolled.Outcomes will be measured at delivery time.

SECONDARY OUTCOMES:
Changing of maternal mean calcium level | 12-14 weeks

OTHER OUTCOMES:
maternal weight gain | 12-14 weeks
neonatal serum calcium level | 12-14 weeks
neonatal growth indices | 12-14 weeks
  neonatal growth indices include neonatal weight, head circumference, length

CONTACTS AND LOCATIONS:
Locations (1):
- Qazvin university of medical science, Kosar hospital, Qazvin, Qazvin Province, Iran

REFERENCES:
- [Derived] Palacios C, Kostiuk LL, Cuthbert A, Weeks J. Vitamin D supplementation for women during pregnancy. Cochrane Database Syst Rev. 2024 Jul 30;7(7):CD008873. doi: 10.1002/14651858.CD008873.pub5. PMID 39077939